CLINICAL TRIAL: NCT01026376
Title: An Expanded Access Program for Decitabine in Patients With Myelodysplastic Syndrome (MDS)
Status: No longer available | Type: Expanded Access
Sponsor: Janssen-Cilag Farmaceutica Ltda. (Industry)
Collaborators: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR015037; DACOGENMYE3001 (Other: Janssen-Cilag Farmaceutica Ltda.)
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes; Decitabine
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine

INTERVENTIONS:
Drug: decitabine — Cycles of 15mg/m2 infusion during 3h, 3 times a day, per 3 days
Drug: decitabine — Cycles of 20mg/m2 infusion during 1h, once a day, per 5 days

SUMMARY:
The purpose of this study is to provide Decitabine to patients with Myelodysplastic syndrome (MDS) of all FAB (French-American-British) subtypes and Intermediate-1, Intermediate-2, and High-Risk International Prognostic Scoring System groups, including both previously treated and untreated patients.

DETAILED DESCRIPTION:
Myelodysplastic Syndromes (MDS), which includes a diverse group of bone marrow disorders that result in ineffective production of blood cells, frequently occurs in elderly patients. Historically, the available treatments for MDS have been symptomatic and supportive, and have not been shown to be effective in producing sustained improvement in hematopoiesis (production of all types of blood cells ) or in delaying leukemic evolution (leukemia is a serious disease in which too many white blood cells are produced, causing weakness and sometimes death). This project is an open-label (all people involved know the identity of the intervention), multicenter, international single arm, Phase 3b study to provide expanded access to Decitabine for patients with myelodysplastic syndromes (MDS). The purpose of this study is to provide Decitabine to patients with Myelodysplastic syndrome (MDS) according some medical classifications: FAB (French-American-British) subtypes and Intermediate-1, Intermediate-2, and High-Risk International Prognostic Scoring System groups, including previously treated and untreated for MDS. The secondary objectives are to evaluate the safety and tolerability of Decitabine, as well as the overall response rate according to the International Working Group (IWG) 2000 and IWG 2006 response criteria, hematologic improvement, cytogenetic response rates (evaluation based on genetic), time to acute myeloid leukemia progression or death (evaluate the length of time that passes prior to onset of leukemia progression and/or death), blood product transfusion requirements per patient (with corresponding dates to collect the number of transfusion independent days), days in the hospital (including reason for hospitalization and the ward within the hospital where the hospitalizations occur) and, optionally, quality of life assessment (EORTC QLQ C-30). 3-day cycle: Decitabine will be administered as a 15mg/m2 administered by continuous infusion over 3 hours repeated every 8 hours for 3 days. 5-day cycle: Another optional schedule could be adopted (at discretion of investigators), Decitabine at a dose of 20mg/m² administered intravenously over 1 hour, once daily for 5 consecutive days, of a 4-week cycle. Treatment may be continued as long as the patient continues to benefit.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of MDS (de novo / primary or secondary) of all FAB subtypes and Intermediate-1, Intermediate-2, and High-Risk International Prognostic Scoring System groups
* Has an Eastern Oncology Cooperative Group (ECOG) performance status of 0-2
* Adequate hepatic and renal function as measured by the following pre-treatment laboratory criteria within 21 days of starting treatment with Decitabine (laboratory measure of liver function no more than 2.5 times the upper limit of normal, laboratory measure of total bilirubin and serum creatinine no more than 1.5 times the upper limit of normal)
* Female patients must be postmenopausal, or surgically sterile, or abstinent, or, if sexually active, be practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study
* Have a negative serum or urine pregnancy test at screening
* Male subjects should be advised not father a child while on or within 2 months of completion of Decitabine therapy

Exclusion Criteria:

* Have a diagnosis of AML (>20% bone marrow blasts) or other progressive malignant disease
* has previously been treated with Azacitidine or Decitabine
* Have uncontrolled heart disease or uncontrolled congestive heart failure
* Have uncontrolled restrictive or obstructive pulmonary disease
* Have active viral or bacterial infection
* Have known positive serology for HIV
* Have a mental illness or any other condition that could prevent full cooperation with the treatment and monitoring requirements of the study
* Have known hypersensitivity to any of the excipients of decitabine
* Are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2008-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Farmaceutica Ltda. Clinical Trial, Study Director — Janssen-Cilag Farmaceutica Ltda.
Locations (11):
- Brazil (9):
  - Belo Horizonte
  - Botucatu
  - Brasília
  - Campinas
  - Fortaleza
  - Pinheiros
  - Rio de Janeiro
  - São Paulo
  - São Paulol
- Hong Kong, Hong Kong
- Bangkok, Thailand